CLINICAL TRIAL: NCT01685840
Title: Guiding Evidence Based Therapy Using Biomarker Intensified Treatment in Heart Failure.
Brief Title: Guiding Evidence Based Therapy Using Biomarker Intensified Treatment
Acronym: GUIDE-IT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Project was stopped due to futility
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00033097
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Experimental): Usual Care group will receive standard heart failure treatment based on the doctor's best judgment and following the recommendation of current guidelines. This will typically include the use of medicines such as beta-blockers, ACE-inhibitors, and diuretics, all of which are approved, recommended treatments for heart failure.
  Interventions: Other: Usual Care
- Biomarker-Guided Care (Experimental): Device: Biomarker-Guided care NT-proBNP The Biomarker Guided Therapy group will receive the standard heart failure treatments. In addition, the doctor will use the results of a blood test called NT-proBNP to help adjust the treatments and drug doses.
  Interventions: Device: Biomarker-guided care NT-proBNP

INTERVENTIONS:
Other: Usual Care — Usual Care
  Arms: Usual Care
Device: Biomarker-guided care NT-proBNP — Device: NT-proBNP
  Arms: Biomarker-Guided Care

SUMMARY:
The primary objective is to determine the efficacy of a strategy of biomarker-guided therapy compared with usual care in high risk patients with left ventricular systolic dysfunction.

DETAILED DESCRIPTION:
Heart failure is a common disorder in which the heart cannot pump enough blood to meet the needs of the rest of the body. Common symptoms of heart failure include shortness of breath, swelling, and fatigue. Standard treatment for heart failure include diuretics to control fluid, as well as drugs called "neurohormonal antagonists" (such as beta-blockers and ACE-inhibitors) that help the heart work more efficiently and prevent worsening of heart function. Typically, doctors adjust these medicines based on their clinical judgment about what doses and combination will work best for you. We are testing whether the use of a blood test called NT-proBNP (which measures a hormone released by the heart) can help doctors do a better job of adjusting these heart failure medicines over time than clinical judgment alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Most recent LVEF to be ≤ 40% by any method within 12 months of randomization.
* High risk heart failure as defined by the following criteria:

A Heart Failure Event in the prior 12 months, defined as any one of the following:

* HF Hospitalization
* Treatment in the Emergency Department (or equivalent) for Heart Failure
* Outpatient treatment for heart failure with intravenous diuretics

AND

* NT-proBNP greater than 2000 pg/mL or BNP greater than 400 pg/mL at any time during the 30 days prior to randomization
* Willing to provide informed consent

Exclusion Criteria:

* Acute coronary syndrome (clinical diagnosis) or cardiac revascularization procedure within 30 days
* Cardiac resynchronization therapy (CRT) within prior 3 months or current plan to implant CRT device
* Active myocarditis, Hypertrophic obstructive cardiomyopathy, pericarditis, or restrictive cardiomyopathy
* Severe stenotic valvular disease
* Anticipated heart transplantation or ventricular assist device within 12 months
* Chronic inotropic therapy
* Complex congenital heart disease
* End stage renal disease with renal replacement therapy
* Non cardiac terminal illness with expected survival less than 12 months
* Women who are pregnant or planning to become pregnant
* Inability to comply with planned study procedures
* Enrollment or planned enrollment in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 894 (Actual)
Dates: Start 2012-12; Primary Completion 2016-09-20 (Actual); Study Completion 2016-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Felker, MD, Principal Investigator — Duke University
Locations (46):
- United States (40):
  - The Heart Center PC, Huntsville, Alabama
  - Sutter Memorial Hospital, Sacramento, California
  - University of California San Diego Medical Center, San Diego, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Holy Cross Medical Group, Coral Springs, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Emory University, Atlanta, Georgia
  - University Cardiology Associates, LLC, Augusta, Georgia
  - Fox Valley Clinical Research Center, LLC, Aurora, Illinois
  - Krannert Institute of Cardiology, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - Metropolitan Cardiovascular Consultants, Beltsville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Medical Center, Boston, Massachusetts
  - Pentucket Medical Associates, Haverhill, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cardiovascular Associates of the Delaware Valley, Cherry Hill, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Cardiovascular Associates of the Delaware Valley, Sewell, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - Saratoga Cardiology Associates, Saratoga Springs, New York
  - Bronx-Lebanon Hospital Center, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York
  - Albert Einstein University Hospital, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Capitol Area Research, LLC, Camp Hill, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - AnMed Health Medical Center, Anderson, South Carolina
  - University of Texas Southwestern Medical Center Dallas, Dallas, Texas
  - Intermountain Medical Center, Murray, Utah
  - Cardiovascular Associates, Ltd., Chesapeake, Virginia
- Canada (6):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Saint Paul's Hospital, Vancouver, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Michaels Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Augusto SN Jr, Wu Y, Chaikijurajai T, Hazen SL, Tang WHW. Abbreviated Duke Activity Status Index for Risk Stratification in Heart Failure. Am J Cardiol. 2025 Feb 15;237:54-59. doi: 10.1016/j.amjcard.2024.11.029. Epub 2024 Nov 26. PMID 39603580
- [Derived] Fuery MA, Leifer ES, Samsky MD, Sen S, O'Connor CM, Fiuzat M, Ezekowitz J, Pina I, Whellan D, Mark D, Felker GM, Desai NR, Januzzi JL, Ahmad T. Prognostic Impact of Repeated NT-proBNP Measurements in Patients With Heart Failure With Reduced Ejection Fraction. JACC Heart Fail. 2024 Mar;12(3):479-487. doi: 10.1016/j.jchf.2023.11.007. Epub 2023 Dec 20. PMID 38127049
- [Derived] Ezekowitz JA, Alemayehu W, Rathwell S, Grant AD, Fiuzat M, Whellan DJ, Ahmad T, Adams K, Pina IL, Cooper LS, Januzzi JL, Leifer ES, Mark D, O'Connor CM, Felker GM. The influence of comorbidities on achieving an N-terminal pro-b-type natriuretic peptide target: a secondary analysis of the GUIDE-IT trial. ESC Heart Fail. 2022 Feb;9(1):77-86. doi: 10.1002/ehf2.13692. Epub 2021 Nov 16. PMID 34784657
- [Derived] Chouairi F, Fuery MA, Mullan CW, Caraballo C, Sen S, Maulion C, Wilkinson ST, Surti T, McCullough M, Miller PE, Pacor J, Leifer ES, Felker GM, Velazquez EJ, Fiuzat M, O'Connor CM, Januzzi JL, Desai NR, Ahmad T. The Impact of Depression on Outcomes in Patients With Heart Failure and Reduced Ejection Fraction Treated in the GUIDE-IT Trial. J Card Fail. 2021 Dec;27(12):1359-1366. doi: 10.1016/j.cardfail.2021.06.008. Epub 2021 Jun 22. PMID 34166799
- [Derived] Fuery MA, Chouairi F, Januzzi JL, Moe GW, Caraballo C, McCullough M, Miller PE, Reinhardt SW, Clark K, Oseran A, Milner A, Pacor J, Kahn PA, Singh A, Ravindra N, Guha A, Vadlamani L, Kulkarni NS, Fiuzat M, Felker GM, O'Connor CM, Ahmad T, Ezekowitz J, Desai NR. Intercountry Differences in Guideline-Directed Medical Therapy and Outcomes Among Patients With Heart Failure. JACC Heart Fail. 2021 Jul;9(7):497-505. doi: 10.1016/j.jchf.2021.02.011. Epub 2021 May 12. PMID 33992564
- [Derived] Daubert MA, Yow E, Barnhart HX, Pina IL, Ahmad T, Leifer E, Cooper L, Desvigne-Nickens P, Fiuzat M, Adams K, Ezekowitz J, Whellan DJ, Januzzi JL, O'Connor CM, Felker GM. Differences in NT-proBNP Response and Prognosis in Men and Women With Heart Failure With Reduced Ejection Fraction. J Am Heart Assoc. 2021 May 18;10(10):e019712. doi: 10.1161/JAHA.120.019712. Epub 2021 May 6. PMID 33955231
- [Derived] Parcha V, Patel N, Kalra R, Suri SS, Arora G, Wang TJ, Arora P. Obesity and Serial NT-proBNP Levels in Guided Medical Therapy for Heart Failure With Reduced Ejection Fraction: Insights From the GUIDE-IT Trial. J Am Heart Assoc. 2021 Apr 6;10(7):e018689. doi: 10.1161/JAHA.120.018689. Epub 2021 Mar 23. PMID 33754794
- [Derived] Fiuzat M, Ezekowitz J, Alemayehu W, Westerhout CM, Sbolli M, Cani D, Whellan DJ, Ahmad T, Adams K, Pina IL, Patel CB, Anstrom KJ, Cooper LS, Mark D, Leifer ES, Felker GM, Januzzi JL, O'Connor CM. Assessment of Limitations to Optimization of Guideline-Directed Medical Therapy in Heart Failure From the GUIDE-IT Trial: A Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2020 Jul 1;5(7):757-764. doi: 10.1001/jamacardio.2020.0640. PMID 32319999
- [Derived] Januzzi JL Jr, Ahmad T, Mulder H, Coles A, Anstrom KJ, Adams KF, Ezekowitz JA, Fiuzat M, Houston-Miller N, Mark DB, Pina IL, Passmore G, Whellan DJ, Cooper LS, Leifer ES, Desvigne-Nickens P, Felker GM, O'Connor CM. Natriuretic Peptide Response and Outcomes in Chronic Heart Failure With Reduced Ejection Fraction. J Am Coll Cardiol. 2019 Sep 3;74(9):1205-1217. doi: 10.1016/j.jacc.2019.06.055. PMID 31466618
- [Derived] O'Connor C, Fiuzat M, Mulder H, Coles A, Ahmad T, Ezekowitz JA, Adams KF, Pina IL, Anstrom KJ, Cooper LS, Mark DB, Whellan DJ, Januzzi JL Jr, Leifer ES, Felker GM. Clinical factors related to morbidity and mortality in high-risk heart failure patients: the GUIDE-IT predictive model and risk score. Eur J Heart Fail. 2019 Jun;21(6):770-778. doi: 10.1002/ejhf.1450. Epub 2019 Mar 27. PMID 30919549
- [Derived] Daubert MA, Adams K, Yow E, Barnhart HX, Douglas PS, Rimmer S, Norris C, Cooper L, Leifer E, Desvigne-Nickens P, Anstrom K, Fiuzat M, Ezekowitz J, Mark DB, O'Connor CM, Januzzi J, Felker GM. NT-proBNP Goal Achievement Is Associated With Significant Reverse Remodeling and Improved Clinical Outcomes in HFrEF. JACC Heart Fail. 2019 Feb;7(2):158-168. doi: 10.1016/j.jchf.2018.10.014. Epub 2019 Jan 2. PMID 30611722
- [Derived] Mark DB, Cowper PA, Anstrom KJ, Sheng S, Daniels MR, Knight JD, Baloch KN, Davidson-Ray L, Fiuzat M, Januzzi JL Jr, Whellan DJ, Pina IL, Ezekowitz JA, Adams KF, Cooper LS, O'Connor CM, Felker GM. Economic and Quality-of-Life Outcomes of Natriuretic Peptide-Guided Therapy for Heart Failure. J Am Coll Cardiol. 2018 Nov 27;72(21):2551-2562. doi: 10.1016/j.jacc.2018.08.2184. PMID 30466512
- [Derived] Felker GM, Anstrom KJ, Adams KF, Ezekowitz JA, Fiuzat M, Houston-Miller N, Januzzi JL Jr, Mark DB, Pina IL, Passmore G, Whellan DJ, Yang H, Cooper LS, Leifer ES, Desvigne-Nickens P, O'Connor CM. Effect of Natriuretic Peptide-Guided Therapy on Hospitalization or Cardiovascular Mortality in High-Risk Patients With Heart Failure and Reduced Ejection Fraction: A Randomized Clinical Trial. JAMA. 2017 Aug 22;318(8):713-720. doi: 10.1001/jama.2017.10565. PMID 28829876
- [Derived] Felker GM, Ahmad T, Anstrom KJ, Adams KF, Cooper LS, Ezekowitz JA, Fiuzat M, Houston-Miller N, Januzzi JL, Leifer ES, Mark DB, Desvigne-Nickens P, Paynter G, Pina IL, Whellan DJ, O'Connor CM. Rationale and design of the GUIDE-IT study: Guiding Evidence Based Therapy Using Biomarker Intensified Treatment in Heart Failure. JACC Heart Fail. 2014 Oct;2(5):457-65. doi: 10.1016/j.jchf.2014.05.007. Epub 2014 Sep 3. PMID 25194287

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 894 participants were randomized
Period: Overall Study
Arm/Group | Usual Care | Biomarker-Guided Care
Started | 448 | 446
Completed | 119 | 114
Not Completed | 329 | 332
Not completed — Death | 77 | 66
Not completed — Lost to Follow-up | 27 | 25
Not completed — Physician Decision | 3 | 7
Not completed — Withdrawal by Subject | 14 | 17
Not completed — Futility | 197 | 200
Not completed — Had VAD, Dialysis or Transplant | 11 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Biomarker-Guided Care | Total
Number analyzed (Participants) | 448 | 446 | 894
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (13.4) | 60.4 (14.3) | 61.5 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 139 | 286
  Male | 301 | 307 | 608
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 30 | 58
  Not Hispanic or Latino | 420 | 416 | 836
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 11 | 16 | 27
  Native Hawaiian or Other Pacific Islander | 3 | 4 | 7
  Black or African American | 155 | 167 | 322
  White | 257 | 228 | 485
  More than one race | 14 | 13 | 27
  Unknown or Not Reported | 7 | 16 | 23

OUTCOME MEASURES:

1. Primary Outcome: CV Death or Heart Failure Hospitalization
Description: Composite of First Heart Failure Hospitalization or Cardiovascular Mortality
Time Frame: 24 Months
Measure: Number; unit: events
Arm/Group | Usual Care | Biomarker-Guided Care
Number analyzed (Participants) | 448 | 446
events | 164 | 164
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-Guided Care; Test type: Superiority or Other; p = 0.88, Regression, Cox — A sample size of 1100 patients was expected to provide approximately 90% power to detect a difference in the primary endpoint with an assumed type I error rate of 0.05, 2-sided. Analysis was adjusted for age, sex, ejection fraction, NT-proBNP and DM; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.79 to 1.22]

2. Secondary Outcome: All-cause Mortality
Description: All-cause mortality by treatment arm
Time Frame: 24 months
Measure: Number; unit: deaths
Arm/Group | Usual Care | Biomarker-Guided Care
Number analyzed (Participants) | 448 | 446
deaths | 77 | 66
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-Guided Care; Test type: Superiority or Other; p = 0.37, Regression, Cox; Cox Proportional Hazard = 0.86, 95% CI 2-sided [0.62 to 1.20]

3. Secondary Outcome: Cumulative Morbidity
Description: Days alive and not hospitalized for CV reasons
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Usual Care | Biomarker-Guided Care
Number analyzed (Participants) | 448 | 446
days | 616 [595 to 637] | 626 [605 to 646]
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-Guided Care; Test type: Superiority or Other; p = 0.53, Bang-Tsiatis Partitioned Estimator; Mean Difference (Net) = 9, 95% CI 2-sided [-20 to 39]

4. Secondary Outcome: CV Death
Description: CV death by treatment arm
Time Frame: 24 months
Measure: Number; unit: deaths
Arm/Group | Usual Care | Biomarker-Guided Care
Number analyzed (Participants) | 448 | 446
deaths | 57 | 53
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-Guided Care; Test type: Superiority or Other; p = 0.75, Regression, Cox; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.65 to 1.37]

5. Secondary Outcome: Number of Hospitalizations for First Heart Failure
Description: First Heart Failure Hospitalization
Time Frame: 24 months
Measure: Number; unit: hospitalizations
Arm/Group | Usual Care | Biomarker-Guided Care
Number analyzed (Participants) | 448 | 446
hospitalizations | 141 | 147
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-Guided Care; Test type: Superiority or Other; p = 0.76, Regression, Cox; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.82 to 1.31]

6. Secondary Outcome: Number of Hospitalizations for Recurrent Heart Failure
Description: Recurrent Heart Failure Hospitalization
Time Frame: 24 months
Measure: Number; unit: hospitalizations
Arm/Group | Usual Care | Biomarker-Guided Care
Number analyzed (Participants) | 448 | 446
hospitalizations | 277 | 350
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-Guided Care; Test type: Superiority or Other; p = 0.08, Anderson-Gill Intensity Model; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.97 to 1.72]

7. Secondary Outcome: Percentage of Patients With Moderate to Severe Depression
Description: Percentage of patients with moderate to severe depression as measured by the Center for Epidemiologic Studies Depression Scale (CES-D).
  CES-D is a 20-item scale measuring general depression. Scores range from 0-60, with higher scores indicating greater general depression. Moderate to severe depression is indicated by a score of 11 or higher.
Time Frame: Baseline, 3,6, 12 and 24 months
Population: "Number of participants analyzed" is the number of participants who completed the questionnaire
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | Biomarker-Guided Care
Number analyzed (Participants) | 439 | 437
percentage of participants
  Baseline | 34.6 | 36.2
  3 month: number analyzed (Participants) | 355 | 345
  3 month | 26.2 | 27.8
  6 month: number analyzed (Participants) | 293 | 301
  6 month | 25.6 | 27.6
  12 month: number analyzed (Participants) | 236 | 254
  12 month | 25.9 | 27.6
  24 month: number analyzed (Participants) | 122 | 132
  24 month | 25.4 | 25.8
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-Guided Care; Baseline; Test type: Superiority; p = 0.636, Mixed Models Analysis
Statistical Analysis 2: Comparison: Usual Care vs Biomarker-Guided Care; 3 month; Test type: Superiority; p = 0.628, Mixed Models Analysis
Statistical Analysis 3: Comparison: Usual Care vs Biomarker-Guided Care; 6 month; Test type: Superiority; p = 0.586, Mixed Models Analysis
Statistical Analysis 4: Comparison: Usual Care vs Biomarker-Guided Care; 12 month; Test type: Superiority; p = 0.669, Mixed Models Analysis
Statistical Analysis 5: Comparison: Usual Care vs Biomarker-Guided Care; 24 month; Test type: Superiority; p = 0.949, Mixed Models Analysis

8. Secondary Outcome: Duke Activity Status Index (DASI)
Description: The DASI is a self-administered questionnaire that measures a patient's functional capacity. It can be used to get a rough estimate of a patient's peak oxygen uptake. The maximum score for the DASI is 58.2 (better functional ability/capacity) and the minimum score is 0 (worse functional ability/capacity).
Time Frame: Baseline, 3, 6, 12 and 24 months
Population: "Number of participants analyzed" is the number of participants who completed the questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Biomarker-Guided Care
Number analyzed (Participants) | 443 | 435
units on a scale
  Baseline | 11.1 (12.6) | 12.6 (13.5)
  3 month: number analyzed (Participants) | 357 | 349
  3 month | 16.9 (14.2) | 17.7 (14.9)
  6 month: number analyzed (Participants) | 298 | 301
  6 month | 17.9 (15.8) | 19.7 (16.6)
  12 month: number analyzed (Participants) | 243 | 260
  12 month | 17.4 (16.1) | 19.3 (17.0)
  24 month: number analyzed (Participants) | 126 | 132
  24 month | 19.6 (17.8) | 18.2 (17.4)
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-Guided Care; 3 month; Test type: Superiority; p = 0.404, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = 0.880, 95% CI 2-sided [-1.188 to 2.947]
Statistical Analysis 2: Comparison: Usual Care vs Biomarker-Guided Care; 6 month; Test type: Superiority; p = 0.219, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = 1.478, 95% CI 2-sided [-0.881 to 3.836]
Statistical Analysis 3: Comparison: Usual Care vs Biomarker-Guided Care; 12 month; Test type: Superiority; p = 0.104, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = 2.099, 95% CI 2-sided [-0.433 to 4.630]
Statistical Analysis 4: Comparison: Usual Care vs Biomarker-Guided Care; 24 month; Test type: Superiority; p = 0.228, Mixed Models Analysis; Mean Difference (Final Values) = 1.999, 95% CI 2-sided [-1.253 to 5.250]

9. Secondary Outcome: EQ-5D Health Index
Description: The EQ-5D measures the subjects health status in 5 categories (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and totals them into 1 score, from -0.59 (worst) to 1 (best).
Time Frame: Baseline, 3, 6, 12 and 24 months
Population: "Number of participants analyzed" is the number of participants who completed the questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Biomarker-Guided Care
Number analyzed (Participants) | 439 | 431
units on a scale
  Baseline | 0.7 (0.3) | 0.7 (0.3)
  3 month: number analyzed (Participants) | 372 | 358
  3 month | 0.7 (0.3) | 0.7 (0.3)
  6 month: number analyzed (Participants) | 319 | 321
  6 month | 0.7 (0.3) | 0.7 (0.3)
  12 month: number analyzed (Participants) | 261 | 269
  12 month | 0.7 (0.3) | 0.7 (0.3)
  24 month: number analyzed (Participants) | 131 | 137
  24 month | 0.7 (0.3) | 0.7 (0.3)
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-Guided Care; 3 month; Test type: Superiority; p = 0.421, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = 0.017, 95% CI 2-sided [-0.025 to 0.060]
Statistical Analysis 2: Comparison: Usual Care vs Biomarker-Guided Care; 6 month; Test type: Superiority; p = 0.239, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = 0.028, 95% CI 2-sided [-0.018 to 0.074]
Statistical Analysis 3: Comparison: Usual Care vs Biomarker-Guided Care; 12 month; Test type: Superiority; p = 0.402, Mixed Models Analysis; Mean Difference (Final Values) = 0.021, 95% CI 2-sided [-0.028 to 0.070]
Statistical Analysis 4: Comparison: Usual Care vs Biomarker-Guided Care; 24 month; Test type: Superiority; p = 0.780, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = 0.009, 95% CI 2-sided [-0.057 to 0.076]

10. Secondary Outcome: EQ-5D Visual Analog Scale
Description: The EQ-5D VAS records participants self-rated health status on a vertical (0-100) scale with higher scores indicating higher Health-Related Quality of Life, where 0 = worst imaginable health state and 100 = best imaginable health state.
Time Frame: Baseline, 3, 6, 12 and 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Biomarker-Guided Care
Number analyzed (Participants) | 446 | 445
units on a scale
  Baseline | 60.2 (37.6) | 59.2 (22.6)
  3 month | 62.3 (25.9) | 60.2 (27.8)
  6 month | 60.5 (26.5) | 61.5 (25.8)
  12 month | 63.7 (25.8) | 62.1 (24.9)
  24 month | 65.9 (24.0) | 60.8 (24.9)
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-Guided Care; 3 month; Test type: Superiority; p = 0.268, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = -2.131, 95% CI 2-sided [-5.902 to 1.640]
Statistical Analysis 2: Comparison: Usual Care vs Biomarker-Guided Care; 6 month; Test type: Superiority; p = 0.599, Mixed Models Analysis; Mean Difference (Final Values) = 1.069, 95% CI 2-sided [-2.921 to 5.058]
Statistical Analysis 3: Comparison: Usual Care vs Biomarker-Guided Care; 12 month; Test type: Superiority; p = 0.852, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = -0.389, 95% CI 2-sided [-4.486 to 3.707]
Statistical Analysis 4: Comparison: Usual Care vs Biomarker-Guided Care; 24 month; Test type: Superiority; p = 0.221, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = -3.343, 95% CI 2-sided [-8.708 to 2.022]

11. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Score
Description: This KCCQ overall score represents the mean of the following 4 scores: Physical Limitation, Total Symptom, Quality of Life, and Social Limitation. Mean scores are transformed to a 0-100 scale with high scores representing better outcomes.
Time Frame: Baseline, 3, 6,12 and 24 months
Population: "Number of participants analyzed" is the number of participants who completed the questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Biomarker-Guided Care
Number analyzed (Participants) | 444 | 441
units on a scale
  Baseline | 57.7 (22.4) | 57.5 (21.6)
  3 month: number analyzed (Participants) | 384 | 373
  3 month | 69.2 (22.8) | 68.8 (22.6)
  6 month: number analyzed (Participants) | 327 | 332
  6 month | 70.1 (22.2) | 70.4 (21.8)
  12 month: number analyzed (Participants) | 270 | 279
  12 month | 70.3 (21.9) | 68.4 (24.3)
  24 month: number analyzed (Participants) | 135 | 143
  24 month | 71.6 (24.4) | 70.2 (22.6)
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-Guided Care; 3 month; Test type: Superiority; p = 0.615, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = -0.816, 95% CI 2-sided [-3.999 to 2.367]
Statistical Analysis 2: Comparison: Usual Care vs Biomarker-Guided Care; 6 month; Test type: Superiority; p = 0.878, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = 0.252, 95% CI 2-sided [-2.977 to 3.482]
Statistical Analysis 3: Comparison: Usual Care vs Biomarker-Guided Care; 12 month; Test type: Superiority; p = 0.441, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = -1.406, 95% CI 2-sided [-4.989 to 2.178]
Statistical Analysis 4: Comparison: Usual Care vs Biomarker-Guided Care; 24 month; Test type: Superiority; p = 0.653, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = 1.091, 95% CI 2-sided [-3.673 to 5.856]

12. Secondary Outcome: Short Form-36 (SF-36) General Health Subscale
Description: SF-36 measures perceived Quality of Life. The following subscales were used: General Health, Mental Health, Social Functioning, Physiological Functioning, and Vitality Each subscale is scored from 0-100 with 0 indicating lowest quality of life.
Time Frame: Baseline, 3, 6, 12 and 24 months
Population: "Number of participants analyzed" is the number of participants who completed the questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Biomarker-Guided Care
Number analyzed (Participants) | 441 | 436
units on a scale
  Baseline | 48.4 (11.1) | 48.6 (10.7)
  3 month: number analyzed (Participants) | 348 | 336
  3 month | 51.1 (12.6) | 50.0 (12.9)
  6 month: number analyzed (Participants) | 287 | 294
  6 month | 50.5 (12.7) | 49.9 (12.9)
  12 month: number analyzed (Participants) | 238 | 250
  12 month | 51.0 (12.2) | 50.8 (12.6)
  24 month: number analyzed (Participants) | 121 | 129
  24 month | 48.8 (12.8) | 50.4 (11.9)
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-Guided Care; 3 month; Test type: Superiority; p = 0.199, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = -1.226, 95% CI 2-sided [-3.097 to 0.645]
Statistical Analysis 2: Comparison: Usual Care vs Biomarker-Guided Care; 6 month; Test type: Superiority; p = 0.465, Mixed Models Analysis; Mean Difference (Final Values) = -0.742, 95% CI 2-sided [-2.735 to 1.250]
Statistical Analysis 3: Comparison: Usual Care vs Biomarker-Guided Care; 12 month; Test type: Superiority; p = 0.943, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = -0.074, 95% CI 2-sided [-2.119 to 1.970]
Statistical Analysis 4: Comparison: Usual Care vs Biomarker-Guided Care; 24 month; Test type: Superiority; p = 0.294, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = 1.478, 95% CI 2-sided [-1.286 to 4.241]

13. Secondary Outcome: Short Form-36 (SF-36) Mental Health Subscale
Description: as for outcome 12
Time Frame: Baseline, 3, 6, 12 and 24 months
Population: "Number of participants analyzed" is the number of participants who completed the questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Biomarker-Guided Care
Number analyzed (Participants) | 441 | 438
units on a scale
  Baseline | 69.7 (20.4) | 69.8 (20.9)
  3 month: number analyzed (Participants) | 352 | 339
  3 month | 77.6 (19.9) | 76.1 (21.5)
  6 month: number analyzed (Participants) | 291 | 298
  6 month | 77.7 (20.5) | 77.1 (21.3)
  12 month: number analyzed (Participants) | 233 | 250
  12 month | 77.5 (20.3) | 76.2 (22.2)
  24 month: number analyzed (Participants) | 122 | 129
  24 month | 79.6 (17.6) | 76.6 (22.1)
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-Guided Care; 3 month; Test type: Superiority; p = 0.294, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = -1.579, 95% CI 2-sided [-4.527 to 1.369]
Statistical Analysis 2: Comparison: Usual Care vs Biomarker-Guided Care; 6 month; Test type: Superiority; p = 0.555, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = -0.946, 95% CI 2-sided [-4.096 to 2.203]
Statistical Analysis 3: Comparison: Usual Care vs Biomarker-Guided Care; 12 month; Test type: Superiority; p = 0.643, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = -0.798, 95% CI 2-sided [-4.178 to 2.583]
Statistical Analysis 4: Comparison: Usual Care vs Biomarker-Guided Care; 24 month; Test type: Superiority; p = 0.757, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = -0.647, 95% CI 2-sided [-4.767 to 3.472]

14. Secondary Outcome: Short Form-36 (SF-36) Social Functioning Subscale
Description: as for outcome 12
Time Frame: Baseline, 3, 6, 12 and 24 months
Population: "Number of participants analyzed" is the number of participants who completed the questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Biomarker-Guided Care
Number analyzed (Participants) | 440 | 437
units on a scale
  Baseline | 60.2 (32.7) | 64.8 (30.1)
  3 month | 75.4 (30.8) | 74.9 (31.8)
  6 month | 77.0 (32.3) | 75.0 (32.1)
  12 month | 76.4 (30.9) | 74.5 (31.5)
  24 month | 76.7 (30.3) | 77.2 (31.7)
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-Guided Care; 3 month; Test type: Superiority; p = 0.837, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = -0.484, 95% CI 2-sided [-5.102 to 4.133]
Statistical Analysis 2: Comparison: Usual Care vs Biomarker-Guided Care; 6 month; Test type: Superiority; p = 0.288, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = -2.693, 95% CI 2-sided [-7.662 to 2.276]
Statistical Analysis 3: Comparison: Usual Care vs Biomarker-Guided Care; 12 month; Test type: Superiority; p = 0.567, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = -1.539, 95% CI 2-sided [-6.810 to 3.732]
Statistical Analysis 4: Comparison: Usual Care vs Biomarker-Guided Care; 24 month; Test type: Superiority; p = 0.475, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = 2.512, 95% CI 2-sided [-4.394 to 9.419]

15. Secondary Outcome: Short Form-36 (SF-36) Physiological Functioning Subscale
Description: as for outcome 12
Time Frame: Baseline, 3, 6, 12 and 24 months
Population: "Number of participants analyzed" is the number of participants who completed the questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Biomarker-Guided Care
Number analyzed (Participants) | 442 | 433
units on a scale
  Baseline | 30.6 (32.1) | 31.5 (31.2)
  3 month: number analyzed (Participants) | 355 | 343
  3 month | 43.5 (35.9) | 43.3 (37.5)
  6 month: number analyzed (Participants) | 294 | 302
  6 month | 43.4 (37.4) | 45.6 (37.2)
  12 month: number analyzed (Participants) | 238 | 253
  12 month | 41.9 (38.2) | 47.4 (37.1)
  24 month: number analyzed (Participants) | 123 | 129
  24 month | 47.0 (38.1) | 43.2 (38.6)
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-Guided Care; 3 month; Test type: Superiority; p = 0.696, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = 1.057, 95% CI 2-sided [-4.250 to 6.364]
Statistical Analysis 2: Comparison: Usual Care vs Biomarker-Guided Care; 6 months; Test type: Superiority; p = 0.497, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = 1.966, 95% CI 2-sided [-3.715 to 7.647]
Statistical Analysis 3: Comparison: Usual Care vs Biomarker-Guided Care; 12 month; Test type: Superiority; p = 0.035, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = 6.564, 95% CI 2-sided [0.456 to 12.673]
Statistical Analysis 4: Comparison: Usual Care vs Biomarker-Guided Care; 24 month; Test type: Superiority; p = 0.488, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = 2.857, 95% CI 2-sided [-5.247 to 10.961]

16. Secondary Outcome: Short Form-36 (SF-36) Vitality Subscale
Description: as for outcome 12
Time Frame: Baseline, 3, 6, 12 and 24 months
Population: "Number of participants analyzed" is the number of participants who completed the questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Biomarker-Guided Care
Number analyzed (Participants) | 441 | 438
units on a scale
  Baseline | 43.9 (22.5) | 44.3 (22.3)
  3 month: number analyzed (Participants) | 353 | 339
  3 month | 54.5 (23.6) | 54.6 (23.6)
  6 month: number analyzed (Participants) | 291 | 296
  6 month | 55.1 (24.6) | 55.8 (23.9)
  12 month: number analyzed (Participants) | 234 | 250
  12 month | 54.4 (23.6) | 55.2 (24.3)
  24 month: number analyzed (Participants) | 123 | 129
  24 month | 57.9 (24.8) | 55.9 (24.2)
Statistical Analysis 1: Comparison: Usual Care vs Biomarker-Guided Care; 3 month; Test type: Superiority; p = 0.992, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = 0.017, 95% CI 2-sided [-3.383 to 3.417]
Statistical Analysis 2: Comparison: Usual Care vs Biomarker-Guided Care; 6 month; Test type: Superiority; p = 0.882, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = 0.280, 95% CI 2-sided [-3.409 to 3.969]
Statistical Analysis 3: Comparison: Usual Care vs Biomarker-Guided Care; 12 month; Test type: Superiority; p = 0.647, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = 0.904, 95% CI 2-sided [-2.973 to 4.782]
Statistical Analysis 4: Comparison: Usual Care vs Biomarker-Guided Care; 24 month; Test type: Superiority; p = 0.903, Mixed Models Analysis — Adjusted P-value; Mean Difference (Final Values) = 0.322, 95% CI 2-sided [-4.894 to 5.538]

17. Secondary Outcome: Resource Utilization
Description: Observed Resource Use
Time Frame: 24 months
Population: US Patients in Economics Substudy
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Biomarker-Guided Care | Usual Care
Number analyzed (Participants) | 373 | 362
events
  Number of Hospitalizations | 1.93 (2.80) | 1.83 (2.36)
  Number of ER only events | 0.57 (1.28) | 0.56 (1.29)
  Number of Rehab facilities | 0.06 (0.35) | 0.06 (0.25)
  Total admissions | 2.56 (3.64) | 2.45 (3.20)
Statistical Analysis 1: Comparison: Biomarker-Guided Care vs Usual Care; Hospitalizations; Test type: Superiority; p = 0.74, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Biomarker-Guided Care vs Usual Care; ER only events; Test type: Superiority; p = 0.45, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Biomarker-Guided Care vs Usual Care; Rehab facilities; Test type: Superiority; p = 0.67, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Biomarker-Guided Care vs Usual Care; Total admissions; Test type: Superiority; p = 0.47, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Resource Utilization Cost
Description: Observed Hospital-Based Cost.
Time Frame: 24 months
Population: US Patients with billing data
Measure: Mean (Standard Deviation); unit: 2016 US dollars
Arm/Group | Biomarker-Guided Care | Usual Care
Number analyzed (Participants) | 363 | 350
2016 US dollars
  Hospital Costs | 47,055 (92,270) | 34,396 (60,842)
  Physician Fees | 2,291 (4,128) | 1,761 (2,601)
  Total Cost | 49,346 (96,082) | 36,157 (63,110)
Statistical Analysis 1: Comparison: Biomarker-Guided Care vs Usual Care; Hospital Costs; Test type: Superiority; p = 0.88, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Biomarker-Guided Care vs Usual Care; Physician Fees; Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Biomarker-Guided Care; Total Cost; Test type: Superiority; p = 0.88, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Randomization through completion of the final study visit at 24 months
Description: SAEs and AEs of Interest that occur from randomization through completion of the final study visit will be reported.
Arm/Group | Usual Care | Biomarker-Guided Care
All-Cause Mortality (participants affected / at risk) | 77/448 | 66/446
Serious Adverse Events (participants affected / at risk) | 36/448 | 51/446
Other Adverse Events (participants affected / at risk) | 157/448 | 178/446
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=448) | Biomarker-Guided Care (N=446)
Symptomatic Hypotension (Cardiac disorders) | 2 | 7
Symptomatic Bradycardia (Cardiac disorders) | 0 | 0
Hyperkalemia (Blood and lymphatic system disorders) | 6 | 11
Worsening renal function (Renal and urinary disorders) | 9 | 16
Other Adverse Events (Investigations) | 19 | 17 — Other Adverse Events
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=448) | Biomarker-Guided Care (N=446)
Symptomatic Hypotension (Cardiac disorders) | 30 | 37
Symptomatic Bradycardia (Cardiac disorders) | 3 | 2
Hyperkalemia (Blood and lymphatic system disorders) | 22 | 30
Worsening renal function (Renal and urinary disorders) | 83 | 91
Other Adverse Events (Investigations) | 19 | 18 — Other Adverse Events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No